CLINICAL TRIAL: NCT06661863
Title: Effectiveness of Autologous Bone and Bioactive Glass for Alveolar Preservation in Alveoli With Infectious Process
Brief Title: Effectiveness of Alveolar Bone Preservation in Alveoli With Infectious Process
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Especialidades Espiritu Santo (Other)
Responsible Party: Principal Investigator, Antonio Lanata Flores, Assistant Professor, Universidad de Especialidades Espiritu Santo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024-ODONT-002C
Record Dates: First submitted 2024-09-03; First posted 2024-10-28 (Actual); Last update posted 2024-10-28 (Actual); Status verified 2024-10

CONDITIONS: Alveolar Bone Loss
Keywords: Alveolar Resorption; Alveolar process; Bone Substitutes; Alveolar Bone Grafting
MeSH Terms: conditions — Alveolar Bone Loss

STUDY DESIGN:
Intervention Model Description: The study includes 28 patients who have a tooth extraction indicated in reference to g. avila-ortiz et al. 2020. They will be divided into 2 randomized groups, 14 sockets with an infectious process will be preserved with autologous bone and the remaining 14 with 58s bioactive glass
Who Masked: Participant
Masking Description: The participants will not know wich biomaterial will be grafted
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- autologous bone (Active Comparator): An autologous bone graft is defined as a living tissue capable of promoting bone healing by transferring that tissue from a donor area to a recipient area. It has been defined as the "gold standard" for having the capacity for osteogenesis, osteoinduction, osteoconduction and providing good structural support, showing high biocompatibility and low immunogenicity, however, autologous bone is limited and has greater morbidity due to the collection of autologous bone from the donor site, increased surgical time, greater infection, inflammation, pain and bleeding.
  Interventions: Procedure: alveolar ridge preservation with autologous bone
- Bioactive glass (Experimental): Bioactive glasses (VB) are a group of synthetic ceramics based on silicates coupled with other minerals. Desirable properties of VB include good biocompatibility, osteoconductivity, antimicrobial activity and a porous structure that promotes vascularization
  Interventions: Procedure: alveolar ridge preservation with bioactive glass

INTERVENTIONS:
Procedure: alveolar ridge preservation with bioactive glass — Bioactive glass grafted into alveolar preservation.
  Arms: Bioactive glass
Procedure: alveolar ridge preservation with autologous bone — Autologous bone graft in alveolar ridge preservation.
  Arms: autologous bone

SUMMARY:
Alveolar ridge preservation (ARP) is a surgical technique that aims to minimize the degree of dimensional changes following extraction. In the healing period after extraction, the alveolar bone (AB) undergoes morphological changes during the remodeling process. The changes become evident immediately after tooth extraction, with greater resorption changes observed during the first two months, and these dimensional changes can be observed 1 year after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age
* Patients with indicated tooth extractions
* Patients who have accepted the conditions of the study

Exclusion Criteria:

* Pregnant patients, breastfeeding or using oral contraceptives
* Smoking patients
* Patients with uncontrolled systemic diseases
* History of autoimmune disease
* Previous traumatic extraction
* Patients taking bisphosphonates or anticoagulants
* Patients who are or have undergone chemotherapy and radiotherapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2024-12-15 (Estimated); Study Completion 2029-12-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate bone formation | The evaluation will occur from enrollment through the end of treatment at 12 months. Assessments will be conducted preoperatively, 7 days post-surgery, as well as at 3, 6, and 12 months following the surgery.
  the dimensional bone changes of the preserved at each stage of healing will be analyzed by computer tomography

CONTACTS AND LOCATIONS:
Locations (1):
- Universidadees, Samborondón, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No